CLINICAL TRIAL: NCT02677922
Title: A Phase 1b/2 Open-Label, Randomized Study of 2 Combinations of Isocitrate Dehydrogenase (IDH) Mutant Targeted Therapies Plus Azacitidine: Oral AG-120 Plus Subcutaneous Azacitidine and Oral AG-221 Plus SC Azacitidine in Subjects With Newly Diagnosed Acute Myeloid Leukemia Harboring an IDH1 or an IDH2 Mutation, Respectively, Who Are Not Candidates to Receive Intensive Induction Chemotherapy
Brief Title: A Study to Assess the Safety and Efficacy of Two Combinations of Isocitrate Dehydrogenase (IDH) Mutant Targeted Therapies Plus Azacitidine in Participants With Newly Diagnosed Acute Myeloid Leukemia (AML) Harboring IDH Mutations Who Are Not Candidates to Receive Intensive Induction Chemotherapy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG-221-AML-005; 2015-003951-23 (EudraCT Number)
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Results first posted 2022-11-22 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute Myeloid Leukemia; Leukemia; Azacitidine; AG-120; AG-221
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — ivosidenib; Azacitidine; enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AG-120 + Azacitidine (Experimental)
  Interventions: Drug: AG-120; Drug: Azacitidine
- AG-221 + Azacitidine (Experimental)
  Interventions: Drug: Azacitidine; Drug: AG-221
- Azacitidine (Experimental)
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: AG-120 — Specified dose on specified days
  Arms: AG-120 + Azacitidine
Drug: Azacitidine — Specified dose on specified days
Drug: AG-221 — Specified dose on specified days
  Arms: AG-221 + Azacitidine

SUMMARY:
The purpose of this study are

1. to determine the recommended combination dose of AG-120 and AG-221 separately when administered with azacitidine and,
2. to investigate the safety, tolerability, and efficacy of the combinations of AG-120 with azacitidine and AG-221 with azacitidine versus with azacitidine alone in participants with acute myeloid leukemia (AML) with the isocitrate dehydrogenase (IDH) enzyme isoforms 1 or 2 mutations, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, primary (ie, de novo) or secondary (progression of Myelodysplastic syndrome [MDS] or myeloproliferative neoplasms [MPN], or therapy-related) acute myeloid leukemia (AML) according to the WHO classification with ≥ 20% leukemic blasts in the bone marrow
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Agree to serial bone marrow aspirate/biopsies

Exclusion Criteria:

* Suspected or proven to have acute promyelocytic leukemia based on morphology, immunophenotype, molecular assay, or karyotype
* AML secondary to chronic myelogenous leukemia (CML)
* Received a targeted agent against an isocitrate dehydrogenase 1 (IDH1) or isocitrate dehydrogenase 2 (IDH2) mutation
* Has or is suspected of having central nervous system (CNS) leukemia. Evaluation of cerebrospinal fluid is only required if CNS involvement by leukemia is suspected during screening

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2025-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (49):
- United States (9):
  - Local Institution - 105, Duarte, California
  - Local Institution - 107, New Haven, Connecticut
  - Local Institution - 108, Chicago, Illinois
  - Local Institution - 103, Chicago, Illinois
  - Local Institution - 102, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Local Institution - 902, Boston, Massachusetts
  - Local Institution - 106, New York, New York
  - Local Institution - 110, Dallas, Texas
- Australia (3):
  - Local Institution - 178, Adelaide, South Australia
  - Local Institution - 175, Melbourne
  - Local Institution - 177, Perth
- Local Institution - UNK-121, Yvoir, Belgium
- Local Institution - 125, Toronto, Ontario, Canada
- France (7):
  - Local Institution - 205, Lille
  - Local Institution - 206, Marseille
  - Local Institution - 200, Paris
  - Local Institution - 204, Pessac
  - Local Institution - 202, Pierre-Bénite
  - Local Institution - 203, Toulouse
  - Local Institution - 201, Villejuif
- Germany (3):
  - Local Institution - 227, Berlin
  - Local Institution - 230, Dresden
  - Local Institution - 225, Ulm
- Italy (7):
  - Local Institution - 253, Bologna, Emilia-Romagna
  - Local Institution - 252, Florence
  - Local Institution - 256, Genova
  - Local Institution - 251, Orbassano
  - Local Institution - 254, Padua
  - Local Institution - 250, Pesaro
  - Local Institution - 255, Roma
- Local Institution - 277, Utrecht, Netherlands
- Local Institution - 327, Lisbon, Portugal
- South Korea (2):
  - Local Institution - 351, Seoul
  - Local Institution - 350, Seoul
- Spain (7):
  - Local Institution - 379, Barcelona
  - Local Institution - 375, Barcelona
  - Local Institution - 376, Cáceres
  - Local Institution - 378, Madrid
  - Local Institution - 381, Madrid
  - Local Institution - 380, Málaga
  - Local Institution - 377, Valencia
- Local Institution - UNK-52, Gothenburg, Sweden
- Switzerland (2):
  - Local Institution - 403, Basel
  - Local Institution - 401, Zurich
- United Kingdom (4):
  - Local Institution - 429, Birmingham
  - Local Institution - 427, Headington
  - Local Institution - 428, London
  - Local Institution - 430, Sutton (Surrey)

REFERENCES:
- [Derived] Montesinos P, Fathi AT, de Botton S, Stein EM, Zeidan AM, Zhu Y, Prebet T, Vigil CE, Bluemmert I, Yu X, DiNardo CD. Differentiation syndrome associated with treatment with IDH2 inhibitor enasidenib: pooled analysis from clinical trials. Blood Adv. 2024 May 28;8(10):2509-2519. doi: 10.1182/bloodadvances.2023011914. PMID 38507688
- [Derived] Woods A, Norsworthy KJ, Wang X, Vallejo J, Chiu Yuen Chow E, Li RJ, Sun J, Charlab R, Jiang X, Pazdur R, Theoret MR, de Claro RA. FDA Approval Summary: Ivosidenib in Combination with Azacitidine for Treatment of Patients with Newly Diagnosed Acute Myeloid Leukemia with an IDH1 Mutation. Clin Cancer Res. 2024 Apr 1;30(7):1226-1231. doi: 10.1158/1078-0432.CCR-23-2234. PMID 38010220
- [Derived] DiNardo CD, Schuh AC, Stein EM, Montesinos P, Wei AH, de Botton S, Zeidan AM, Fathi AT, Kantarjian HM, Bennett JM, Frattini MG, Martin-Regueira P, Lersch F, Gong J, Hasan M, Vyas P, Dohner H. Enasidenib plus azacitidine versus azacitidine alone in patients with newly diagnosed, mutant-IDH2 acute myeloid leukaemia (AG221-AML-005): a single-arm, phase 1b and randomised, phase 2 trial. Lancet Oncol. 2021 Nov;22(11):1597-1608. doi: 10.1016/S1470-2045(21)00494-0. Epub 2021 Oct 18. PMID 34672961
- [Derived] DiNardo CD, Stein AS, Stein EM, Fathi AT, Frankfurt O, Schuh AC, Dohner H, Martinelli G, Patel PA, Raffoux E, Tan P, Zeidan AM, de Botton S, Kantarjian HM, Stone RM, Frattini MG, Lersch F, Gong J, Gianolio DA, Zhang V, Franovic A, Fan B, Goldwasser M, Daigle S, Choe S, Wu B, Winkler T, Vyas P. Mutant Isocitrate Dehydrogenase 1 Inhibitor Ivosidenib in Combination With Azacitidine for Newly Diagnosed Acute Myeloid Leukemia. J Clin Oncol. 2021 Jan 1;39(1):57-65. doi: 10.1200/JCO.20.01632. Epub 2020 Oct 29. PMID 33119479
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA: Participants with an IDH2 mutation receive Azacitidine SC 75 mg/m2/day for 7 days of every 28-day treatment cycle was co-administered with AG-221 tablets given at 100 mg orally QD on Days 1 to 28 of each 28-day cycle.
- Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA: Participants with an IDH2 mutation receive Azacitidine SC 75 mg/m2/day for 7 days of every 28-day treatment cycle was co-administered with AG-221 tablets given at 200 mg, orally QD on Days 1 to 28 of each 28-day cycle.
- Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA: Participants with an IDH1 mutation receive Azacitidine SC 75 mg/m2/day for 7 days of every 28-day treatment cycle was co-administered with AG-120 tablets given at 500 mg orally once a day (QD) on Days 1 to 28 of each 28-day cycle.
- Phase 1b Expansion Stage: AG-120 (500mg) + AZA: Participants with an IDH1 mutation receive Azacitidine SC 75 mg/m2/day for 7 days of every 28-day treatment cycle was co-administered with AG-120 tablets was given at 500 mg orally once a day (QD) on Days 1 to 28 of each 28-day cycle.
- Phase 2 Randomized Stage: AG-221 (100mg) + AZA: Azacitidine SC 75 mg/m2/day for 7 days of every 28-day treatment cycle was co-administered with AG-221 tablets given at 100mg orally once a day (QD) on Days 1 to 28 of each 28-day cycle.
- Phase 2 Randomized Stage: AZA Monotherapy: Azacitidine monotherapy was administered SC at 75 mg/m2/day for 7 days of every 28-day treatment cycle
Period: Pre-Treatment Period
Arm/Group | Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA | Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA | Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA | Phase 1b Expansion Stage: AG-120 (500mg) + AZA | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Started | 3 | 3 | 7 | 16 | 68 | 33
Completed | 3 | 3 | 7 | 16 | 68 | 32
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period
Arm/Group | Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA | Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA | Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA | Phase 1b Expansion Stage: AG-120 (500mg) + AZA | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Started | 3 | 3 | 7 | 16 | 68 | 32
Completed (Ongoing) | 1 | 1 | 4 | 3 | 21 | 1
Not Completed | 2 | 2 | 3 | 13 | 47 | 31
Not completed — Adverse Event | 0 | 0 | 1 | 3 | 5 | 2
Not completed — Progressive Disease | 1 | 1 | 0 | 0 | 8 | 7
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 1 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3 | 5 | 5
Not completed — Transition to Commercially Available Treatment | 0 | 1 | 1 | 1 | 1 | 2
Not completed — Disease Relapse | 0 | 0 | 0 | 3 | 6 | 1
Not completed — Allogeneic HSCT | 1 | 0 | 0 | 1 | 4 | 1
Not completed — Other Reasons | 0 | 0 | 0 | 1 | 3 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 12 | 1
Not completed — Non-compliance with Study Drug | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA | Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA | Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA | Phase 1b Expansion Stage: AG-120 (500mg) + AZA | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy | Total
Number analyzed (Participants) | 3 | 3 | 7 | 16 | 68 | 33 | 130
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 0 | 1 | 0 | 3 | 7 | 1 | 12
  >= 65-< 75 | 1 | 2 | 2 | 6 | 22 | 14 | 47
  >= 75 | 2 | 0 | 5 | 7 | 39 | 18 | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 9 | 36 | 11 | 63
  Male | 1 | 1 | 4 | 7 | 32 | 22 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 3 | 3 | 6 | 14 | 51 | 26 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 16 | 6 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 5 | 1 | 8
  White | 2 | 2 | 7 | 13 | 49 | 24 | 97
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 13 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing Dose-limiting Toxicities (DLTs): Phase 1B (Dose Finding Stage)
Description: Dose-limiting toxicities (DLTs) are defined as an event that constitute a change from baseline irrespective of outcome and determined by the investigator to be related to treatment. The DLT-evaluable participants were defined as participants who took at least 1 dose of study drug in the Phase 1b Dose-Finding Stage and either had a DLT during Cycle 1 (regardless of amount of study drug exposure), or had no DLT and completed at least 75% of AG-120 or AG-221 doses (21 out of 28 days) and a minimum of 5 doses of AZA, at least 50% of the planned combination doses for AG-120 or AG-221 and AZA administered together (in the same day for 4 out of 7 days) in the first 28 days from C1D1, and were also considered by the Clinical Study Team to have sufficient safety data available to conclude that a DLT did not occur during Cycle 1.
Time Frame: From first dose to 28 days after first dose
Population: All DLT evaluable participants in the Phase 1b (Dose-finding Stage)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA | Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA | Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA
Number analyzed (Participants) | 3 | 3 | 7
Participants | 0 | 0 | 0

2. Primary Outcome: The Number of Participants Experiencing Adverse Events: Phase 1B (Dose Finding and Expansion Stage)
Description: The number of participants experiencing different types of adverse events (AE). An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. A Serious Adverse Event (SAE) is any AE occurring at any dose that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, and/or constitutes an important medical event. Adverse events were analyzed in terms of treatment-emergent AEs (TEAEs). Treatment-emergent adverse events (TEAE) was defined as events that began on or after the start of study drug through 28 days after the last study treatment. The severity/intensity of AEs were graded based upon the Common Terminology Criteria for Adverse Events (CTCAE, Version 4.03) where Grade 3 = Severe, Grade 4 = Life-threatening, and Grade 5 = Death.
Time Frame: From first dose to 28 days after last dose (up to approximately 13 months)
Population: All treated participants in Phase 1B (Dose Finding and Expansion Stage)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA | Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA | Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA | Phase 1b Expansion Stage: AG-120 (500mg) + AZA
Number analyzed (Participants) | 3 | 3 | 7 | 16
Participants
  Participants with at Least One TEAE | 3 | 3 | 7 | 16
  Participants with at Least One TEAE Related to Study Drug(s) | 3 | 3 | 7 | 16
  Participants with at Least One Grade 3-4 TEAE | 3 | 3 | 7 | 15
  Participants with at least One Grade 3-4 TEAE Related to Study Drug(s) | 2 | 2 | 4 | 10
  Participants with at Least One Grade 5 TEAE | 0 | 1 | 1 | 2
  Participants with at Least One Grade 5 TEAE Related to Study Drug(s) | 0 | 0 | 0 | 0
  Participants with at Least One Serious TEAE | 3 | 2 | 4 | 11
  Participants with at Least One Serious TEAE Related to Study Drug(s) | 0 | 1 | 1 | 5
  Participants with at Least One TEAE Leading to Discontinuation of Study Drug(s) | 1 | 0 | 1 | 4
  Participants with at Least One Study Drug Related TEAE Leading to Discontinuation of Study Drug | 0 | 0 | 0 | 1
  Participants with at Least One TEAE Leading to Dose Reduction of Study Drug(s) | 1 | 1 | 2 | 5
  Participants with at Least One TEAE Leading to Dose Interruption of Study Drug(s) | 3 | 3 | 2 | 11
  Participants with at Least One Study Drug(s) Related TEAE Leading to Study Drug Dose Reduction | 0 | 1 | 1 | 5
  Participants with at Least One Study Drug(s) Related TEAE Leading to Study Drug Dose Interruption | 1 | 2 | 2 | 8

3. Primary Outcome: Overall Response Rate: Phase 2 (Randomized Stage)
Description: The percent of participants with MLFS + CR + CRi + CRp + PR according to modified International Working Group Acute Myeloid Leukemia (IWG AML) response criteria as assessed by investigator. Complete response (CR) and morphologic leukemia-free state (MLFS) are defined as <5% blasts in a BM aspirate sample with marrow spicules and a count of ≥200 nucleated cells. There should be no blasts with Auer rods and no extramedullary disease. CR must also include: absolute neutrophil count (ANC) ≥1,000/μL, Platelet count ≥100,000/μL, and independent of red cell transfusions for ≥1 week before each response assessment. Complete remission with incomplete neutrophil recovery (CRi) is all criteria of CR except ANC. Complete remission with incomplete platelet recovery (CRp) is all criteria of CR except platelet count. Partial remission (PR) is defined as all hematologic criteria of CR with a >50% decrease in the percentage of BM blasts to 5% to 25%. (<5% considered if Auer rods are present).
Time Frame: From first dose up to approximately 26 months
Population: All randomized participants in Phase 2 (Randomized Stage)
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 68 | 33
Percent of Participants | 73.5 [61.4 to 83.5] | 36.4 [20.4 to 54.9]
Statistical Analysis 1: Comparison: Phase 2 Randomized Stage: AG-221 (100mg) + AZA vs Phase 2 Randomized Stage: AZA Monotherapy; Test type: Superiority; p = 0.0003, Chi-squared; Odds Ratio (OR) = 4.86, 95% CI 2-sided [1.99 to 11.85]

4. Secondary Outcome: Overall Response Rate: Phase 1B (Dose Finding and Expansion Stage)
Description: Percent of participants with MLFS + CR + CRi + CRp + PR according to modified International Working Group Acute Myeloid Leukemia (IWG AML) response criteria as assessed by investigator. Complete response (CR) and morphologic leukemia-free state (MLFS) are defined as <5% blasts in a BM aspirate sample with marrow spicules and a count of ≥200 nucleated cells. There should be no blasts with Auer rods and no extramedullary disease. CR must also include: absolute neutrophil count (ANC) ≥1,000/μL, Platelet count ≥100,000/μL, and independent of red cell transfusions for ≥1 week before each response assessment. Complete remission with incomplete neutrophil recovery (CRi) is all criteria of CR except ANC. Complete remission with incomplete platelet recovery (CRp) is all criteria of CR except platelet count. Partial remission (PR) is defined as all hematologic criteria of CR with a >50% decrease in the percentage of BM blasts to 5% to 25%. (<5% considered if Auer rods are present).
Time Frame: From first dose up to approximately 13 months
Population: All treated participants in Phase 1B (Dose Finding and Expansion Stage)
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA | Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA | Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA | Phase 1b Expansion Stage: AG-120 (500mg) + AZA
Number analyzed (Participants) | 3 | 3 | 7 | 16
Percent of Participants | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 100 [59.0 to 100] | 68.8 [41.3 to 89.0]

5. Secondary Outcome: Sponsor Derived CR and CRh: Phase 1B (Dose Finding and Expansion Stage)
Description: The percent of participants with morphologic complete remission (CR) and morphologic complete remission with partial hematologic recovery (CRh) based on laboratory data. CR is defined as less than 5% blasts in a BM aspirate sample with marrow spicules and with a count of at least 200 nucleated cells. There should be no blasts with Auer rods and absence of extramedullary disease. Plus, all the following conditions should be met: ANC ≥ 1 x 109/L (1,000/μL), platelet count ≥ 100 x 109/L (100,000/μL), independent of red cell transfusions for ≥ 1 week immediately before each response assessment. CRh is defined as less than 5% blasts in a BM aspirate sample with marrow spicules plus ANC > 500 x 109/L (1,000/μL) & Platelet count > 50 x 109/L (100,000/μL). CRh is defined as Response of bone marrow blast <5% with absolute neutrophil count (ANC) > 0.5 × 10^9/L and platelet > 50 × 10^9/L.
Time Frame: From first dose up to approximately 13 months
Population: All treated participants in Phase 1B (Dose Finding and Expansion Stage)
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA | Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA | Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA | Phase 1b Expansion Stage: AG-120 (500mg) + AZA
Number analyzed (Participants) | 3 | 3 | 7 | 16
Percent of Participants | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 71.4 [29.0 to 96.3] | 62.5 [35.4 to 84.8]

6. Secondary Outcome: Event-free Survival (EFS): Phase 2 (Randomized Stage)
Description: Event-Free Survival is the time from date of randomization to the date of documented morphologic relapse, progression, or death from any cause, whichever occurs first. Morphologic Relapse is defined as either reappearance of ≥ 5% blasts in the BM not attributable to any other cause or the development of extramedullary disease. Progression is defined as a > 50% increase of BM blast count percentage from baseline to ≥ 20% for participants with 5 to 70% BM blasts at baseline or a doubling of absolute blast count in peripheral blood from baseline to ≥ 10 x 109/L (10,000/μL) for participants with > 70% BM blasts at baseline or the development of new extramedullary disease.
Time Frame: From randomization to the date of documented relapse, progression, or death due to any cause, whichever occurs first (up to approximately 26 months)
Population: All randomized participants in Phase 2 (Randomized Stage)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 68 | 33
Months | 15.9 [13.0 to NA] — Insufficient number of participants with events | 11.9 [8.2 to 15.5]
Statistical Analysis 1: Comparison: Phase 2 Randomized Stage: AG-221 (100mg) + AZA vs Phase 2 Randomized Stage: AZA Monotherapy; Test type: Superiority; p = 0.1083, Log Rank; Cox Proportional Hazard = 0.59, 95% CI 2-sided [0.30 to 1.13]

7. Secondary Outcome: The Number of Participants Experiencing Adverse Events: Phase 2 (Randomized Stage)
Description: as for outcome 2
Time Frame: From first dose to 28 days after last dose (up to approximately 26 months)
Population: All treated participants in Phase 2 (Randomized Stage)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 68 | 32
Participants
  Participants with at Least One TEAE | 68 | 32
  Participants with at Least One TEAE Related to Study Drug(s) | 62 | 26
  Participants with at Least One Grade 3-4 TEAE | 68 | 31
  Participants with at least One Grade 3-4 TEAE Related to Study Drug(s) | 50 | 20
  Participants with at Least One Grade 5 TEAE | 15 | 2
  Participants with at Least One Grade 5 TEAE Related to Study Drug(s) | 0 | 0
  Participants with at Least One Serious TEAE | 64 | 25
  Participants with at Least One Serious TEAE Related to Study Drug(s) | 29 | 14

8. Secondary Outcome: Complete Remission Rate: Phase 2 (Randomized Stage)
Description: The percent of participants with morphologic complete remission (CR) according to modified International Working Group Acute Myeloid Leukemia Response Criteria (IWG AML). CR is defined as less than 5% blasts in a BM aspirate sample with marrow spicules and with a count of at least 200 nucleated cells. There should be no blasts with Auer rods and absence of extramedullary disease; plus the following conditions: absolute neutrophil count (ANC) ≥1,000/μL, Platelet count ≥100,000/μL, and independent of red cell transfusions for ≥1 week before each response assessment.
Time Frame: From first dose up to approximately 26 months
Population: All randomized participants in Phase 2 (Randomized Stage)
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 68 | 33
Percent of Participants | 54.4 [41.9 to 66.5] | 12.1 [3.4 to 28.2]
Statistical Analysis 1: Comparison: Phase 2 Randomized Stage: AG-221 (100mg) + AZA vs Phase 2 Randomized Stage: AZA Monotherapy; Test type: Superiority; p < 0.001, Chi-squared; Odds Ratio (OR) = 8.65, 95% CI 2-sided [2.74 to 27.31]

9. Secondary Outcome: Hematologic Improvement (HI) Rate: Phase 2 (Randomized Stage)
Description: The percent of participants with hematologic improvement neutrophil response (HI-N) + hematologic improvement platelet response (HI-P) + hematologic improvement erythroid response (HI-E) according to the International Working Group for Myelodysplastic Syndromes for Hematologic Improvement (IWG MDS HI) criteria. HI-E is defined as a hemoglobin increase by ≥ 1.5 g/dL and a relevant reduction in units of RBC transfusions by an absolute number of at least 4 RBC transfusions/8 week compared with the pretreatment transfusion number in the previous 8 week. HI-P is defined as an absolute increase of ≥ 30 X 10^9/L for participants starting with > 20 X and an increase from < 20 X 10^9/L to > 20 X 10^9/L and by at least 100%. HI-N is defined as At least 100% increase and an absolute increase > 0.5 X 10^9/L.
Time Frame: From first dose up to approximately 26 months
Population: All randomized participants in Phase 2 (Randomized Stage)
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 68 | 33
Percent of Participants | 70.6 [58.3 to 81.0] | 57.6 [39.2 to 74.5]
Statistical Analysis 1: Comparison: Phase 2 Randomized Stage: AG-221 (100mg) + AZA vs Phase 2 Randomized Stage: AZA Monotherapy; Test type: Superiority; p = 0.1943, Chi-squared; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.74 to 4.20]

10. Secondary Outcome: Duration of Response: Phase 2 (Randomized Stage)
Description: The time from first documented CR/CRi/CRp/PR/MLFS to documented morphologic relapse, progression, or death due to any cause, whichever occurred first. CR and MLFS are defined as <5% blasts in a BM aspirate sample with marrow spicules + a count of ≥200 nucleated cells with no blasts with Auer rods + no extramedullary disease. CR must also include: ANC ≥ 1,000/μL, Platelet count ≥100,000/μL, + independent of red cell transfusions for ≥1 week before assessment. CRi is all criteria of CR except ANC. CRp is all criteria of CR except platelet count. PR is defined as all hematologic criteria of CR with >50% decrease in BM blasts to 5%-25%. Relapse is defined as reappearance of ≥ 5% blasts in the BM not attributable to other cause or development of extramedullary disease. Progression is defined as > 50% increase of BM blast count from baseline to ≥ 20% or a doubling of absolute blast count in peripheral blood from baseline to ≥ 10,000/μL or development of new extramedullary disease.
Time Frame: From first dose up to approximately 26 months
Population: All randomized participants in Phase 2 (Randomized Stage) who achieved CR/CRi/CRp/PR/MLFS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 50 | 12
Months | 24.1 [10.0 to NA] — Insufficient number of participants with events | 9.9 [5.5 to 13.6]

11. Secondary Outcome: Time to Response: Phase 2 (Randomized Stage)
Description: Time from first dose of study drug to first documented MLFS/CR/CRi/CRp/PR according to modified IWG AML response criteria. Complete remission (CR) and morphologic leukemia-free state (MLFS) are defined as <5% blasts in a BM aspirate sample with marrow spicules and a count of ≥200 nucleated cells. There should be no blasts with Auer rods and no extramedullary disease. CR must also include the following conditions: absolute neutrophil count (ANC) ≥1,000/μL, Platelet count ≥100,000/μL, and independent of red cell transfusions for ≥1 week before each response assessment. Complete remission with incomplete neutrophil recovery (CRi) is all criteria of CR except ANC. Complete remission with incomplete platelet recovery (CRp) is all criteria of CR except platelet count. partial remission (PR) is defined as all hematologic criteria of CR with a >50% decrease in the percentage of BM blasts to 5% to 25%. (<5% considered if Auer rods are present).
Time Frame: From first dose to to first documented MLFS/CR/CRi/CRp/PR (up to approximately 26 months)
Population: All randomized participants in Phase 2 (Randomized Stage) who achieved CR/CRi/CRp/PR/MLFS
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 50 | 12
Months | 3.05 (2.551) | 3.42 (1.720)

12. Secondary Outcome: Overall Survival: Phase 2 (Randomized Stage)
Description: Overall survival (OS) is defined as time from randomization to death due to any cause.
Time Frame: From randomization to date of death (up to approximately 26 months)
Population: All randomized participants in Phase 2 (Randomized Stage)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 68 | 33
Months | 22.0 [14.6 to NA] — Insufficient number of participants with events | 22.3 [11.9 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Phase 2 Randomized Stage: AG-221 (100mg) + AZA vs Phase 2 Randomized Stage: AZA Monotherapy; Test type: Superiority; p = 0.9720, Log Rank; Unstratified log-rank test; Cox Proportional Hazard = 0.99, 95% CI 2-sided [0.52 to 1.87] — Cox proportional hazards regression model

13. Secondary Outcome: One Year Survival Rate: Phase 2 (Randomized Stage)
Description: The percent of participants alive at 1 year from randomization
Time Frame: From randomization to 1 year after randomization
Population: All randomized participants in Phase 2 (Randomized Stage)
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 68 | 33
Percent of Participants | 72.2 [59.6 to 81.5] | 69.6 [49.6 to 82.9]
Statistical Analysis 1: Comparison: Phase 2 Randomized Stage: AG-221 (100mg) + AZA vs Phase 2 Randomized Stage: AZA Monotherapy; Test type: Other — Confidence interval of difference; Difference = 2.6, 95% CI 2-sided [-17.3 to 22.5] — The CI for the difference was derived using Greenwood's variance estimate

14. Secondary Outcome: AUC (0-8)- Area Under the Plasma Concentration-Time Curve: Phase 1B (Expansion Stage)
Description: Area under the plasma concentration-time curve from time zero to 8 hours, calculated using the linear trapezoid rule.
Time Frame: Pre-dose, 0.5, 2, 3, 4, 6, 8 hours post dose (± 10 minutes) on day 1 of cycle 1 and 2
Population: All AG-120 treated participants with available pharmacokinetic measurements in Phase 1B (Expansion Stage)
Measure: Mean (Standard Deviation); unit: (h*ng/mL)
Arm/Group | Phase 1b Expansion Stage: AG-120 (500mg) + AZA
Number analyzed (Participants) | 12
(h*ng/mL)
  CYCLE 1 DAY 1 | 31952.4465 (16008.00412)
  CYCLE 2 DAY 1 | 44291.5504 (18806.17037)

15. Secondary Outcome: Cmax- Maximum Observed Plasma Concentration: Phase 1B (Expansion Stage)
Description: Cmax: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data
Time Frame: Pre-dose, 0.5, 2, 3, 4, 6, 8 hours post dose (± 10 minutes) on day 1 of cycle 1 and 2
Population: All AG-120 treated participants with available pharmacokinetic measurements in Phase 1B (Expansion Stage)
Measure: Mean (Standard Deviation); unit: (ng/mL)
Arm/Group | Phase 1b Expansion Stage: AG-120 (500mg) + AZA
Number analyzed (Participants) | 15
(ng/mL)
  CYCLE 1 DAY 1 | 6058.0 (2750.97)
  CYCLE 2 DAY 1: number analyzed (Participants) | 14
  CYCLE 2 DAY 1 | 6340.7 (3191.00)

16. Secondary Outcome: Tmax- Time of Maximum Observed Plasma Concentration: Phase 1B (Expansion Stage)
Description: Tmax: Time of maximum observed plasma concentration, obtained directly from the observed concentration versus time data.
Time Frame: Pre-dose, 0.5, 2, 3, 4, 6, 8 hours post dose (± 10 minutes) on day 1 of cycle 1 and 2
Population: All AG-120 treated participants with available pharmacokinetic measurements in Phase 1B (Expansion Stage)
Measure: Median (Full Range); unit: (h)
Arm/Group | Phase 1b Expansion Stage: AG-120 (500mg) + AZA
Number analyzed (Participants) | 15
(h)
  CYCLE 1 DAY 1 | 3.0000 [0.500 to 8.067]
  CYCLE 2 DAY 1: number analyzed (Participants) | 14
  CYCLE 2 DAY 1 | 2.5000 [0.500 to 7.850]

17. Secondary Outcome: AUC (0-8)- Area Under the Plasma Concentration-Time Curve: Phase 2 (Randomized Stage)
Description: Area under the plasma concentration-time curve from time zero to 8 hours, calculated using the linear trapezoid rule.
Time Frame: Pre-dose, 2, 3, 4, 6, and 8 hours post dose (± 10 minutes) on day 1 of cycle 2
Population: All AG-221 treated participants with available pharmacokinetic measurements in Phase 2 (Randomized Stage)
Measure: Mean (Standard Deviation); unit: (h*ng/mL)
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA
Number analyzed (Participants) | 16
(h*ng/mL) | 100302.8231 (61286.98611)

18. Secondary Outcome: AUC (0-24)- Area Under the Plasma Concentration-Time Curve: Phase 2 (Randomized Stage)
Description: AUC0-24: Area under the plasma concentration-time curve from time zero to 24 hours, calculated using the linear trapezoid rule.
Time Frame: Pre-dose, 2, 3, 4, 6, 8, and 24 hours post dose (± 10 minutes) on day 1 of cycle 2
Population: All AG-221 treated participants with available pharmacokinetic measurements in Phase 2 (Randomized Stage)
Measure: Mean (Standard Deviation); unit: (h*ng/mL)
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA
Number analyzed (Participants) | 13
(h*ng/mL) | 285864.2637 (190300.31922)

19. Secondary Outcome: Cmax- Maximum Observed Plasma Concentration: Phase 2 (Randomized Stage)
Description: Cmax: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data.
Time Frame: Pre-dose, 2, 3, 4, 6, 8, and 24 hours post dose (± 10 minutes) on day 1 of cycle 2
Population: All AG-221 treated participants with available pharmacokinetic measurements in Phase 2 (Randomized Stage)
Measure: Mean (Standard Deviation); unit: (ng/mL)
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA
Number analyzed (Participants) | 16
(ng/mL) | 15965.0 (9663.47)

20. Secondary Outcome: Tmax- Time of Maximum Observed Plasma Concentration: Phase 2 (Randomized Stage)
Description: Tmax: Time of maximum observed plasma concentration, obtained directly from the observed concentration versus time data.
Time Frame: Pre-dose, 2, 3, 4, 6, 8, and 24 hours post dose (± 10 minutes) on day 1 of cycle 2
Population: All AG-221 treated participants with available pharmacokinetic measurements in Phase 2 (Randomized Stage)
Measure: Median (Full Range); unit: (h)
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA
Number analyzed (Participants) | 16
(h) | 2.5333 [0.000 to 23.917]

21. Secondary Outcome: Change From Baseline in Health-related Quality-of-Life Domain Scores of the EORTC QLQ-C30: Phase 2 (Randomized Stage)
Description: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) is composed of 30 items that address general physical symptoms, physical functioning, fatigue and malaise, and social and emotional functioning. Subscale scores are transformed to a 0 to 100 scale, with higher scores on functional scales indicating better function and higher scores on symptom scales indicating worse symptoms. Baseline results are obtained just prior to the start of study treatment on Day 1 of Cycle 1 and will serve as the baseline values. EORTC QLQ-C30 is assessed prior to dosing and prior to interaction with study personnel.
Time Frame: Baseline and Day 1 Cycle 5
Population: All randomized participants with baseline and at least one post-baseline assessment in Phase 2 (Randomized Stage)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 28 | 17
Score on a scale
  Global QoL | 12.2 (27.36) | 4.9 (27.33)
  Physical functioning | 1.9 (20.6) | 6.7 (23.57)
  Role functioning | -0.6 (29.57) | 1.0 (30.88)
  Cognitive functioning | -4.8 (26.00) | 4.9 (25.53)
  Emotional functioning | 7.7 (24.42) | 8.8 (18.51)
  Social functioning | -6.5 (29.52) | 6.9 (34.89)
  Fatigue | -17.5 (33.05) | -8.5 (31.06)
  Nausea and vomiting | -6.0 (29.47) | 1.0 (16.11)
  Pain | -13.1 (33.13) | -4.9 (30.48)
  Dyspnea | -27.4 (35.20) | -9.8 (28.30)
  Insomnia | -6.0 (25.75) | -13.7 (26.51)
  Appetite loss | -7.1 (42.90) | -5.9 (35.81)
  Constipation | 6.0 (32.78) | -9.8 (22.87)
  Diarrhea | -7.1 (31.89) | -5.9 (29.43)
  Financial difficulties | 8.3 (19.51) | -2.0 (34.30)

22. Secondary Outcome: Change From Baseline in Health Utility Indices of the EQ-5D-5L: Phase 2 (Randomized Stage)
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. These health states are converted to a single index value using the crosswalk method to the EQ-5D-3L value set from the United Kingdom (UK). The EQ-5D-3L health utility index based on the UK population weights range from -0.594 to 1.0 with higher scores indicating higher health utility. Baseline results are obtained just prior to the start of study treatment on Day 1 of Cycle 1 and will serve as the baseline values.
Time Frame: Baseline and Day 1 Cycle 5
Population: All randomized participants with baseline and at least one post-baseline assessment in Phase 2 (Randomized Stage)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 28 | 14
Score on a scale | 0.04 (0.216) | 0.02 (0.211)

23. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Scores of the EQ-5D-5L: Phase 2 (Randomized Stage)
Description: The European Quality of Life 5D-5L (EQ-5D-5L) instrument has a respondent's self-rated today's health scale which is recorded on a VAS with endpoints labeled "the best health you can imagine" and "the worst health you can imagine." The scale is numbered from 0 to 100 with 0 corresponding to the worst imaginable health state and 100 corresponding to the best imaginable health state. A high score represents a better level of QoL. Baseline results are obtained just prior to the start of study treatment on Day 1 of Cycle 1 and will serve as the baseline values.
Time Frame: Baseline and Day 1 Cycle 5
Population: All randomized participants with baseline and at least one post-baseline assessment in Phase 2 (Randomized Stage)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
Number analyzed (Participants) | 28 | 17
Score on a scale | 13.00 (26.166) | 1.65 (27.897)

24. Secondary Outcome: Sponsor Derived CR: Phase 2 (Randomized Stage)
Description: The number of participants with Morphologic Complete Remission (CR) based on laboratory data. CR is defined as as less than 5% blasts in a BM aspirate sample with marrow spicules and with a count of at least 200 nucleated cells. There should be no blasts with Auer rods and absence of extramedullary disease. Plus, all the following conditions should be met: ANC ≥ 1 x 109/L (1,000/μL), platelet count ≥ 100 x 109/L (100,000/μL), independent of red cell transfusions for ≥ 1 week immediately before each response assessment.
Time Frame: From first dose to end of study
Reporting Status: Not Posted, anticipated posting 2026-09

25. Secondary Outcome: Sponsor Derived CR and CRh: Phase 2 (Randomized Phase)
Description: The number of participants with morphologic complete remission (CR) and morphologic complete remission with partial hematologic recovery (CRh) based on laboratory data. CR is defined as less than 5% blasts in a BM aspirate sample with marrow spicules and with a count of at least 200 nucleated cells. There should be no blasts with Auer rods and absence of extramedullary disease. Plus, all the following conditions should be met: ANC ≥ 1 x 109/L (1,000/μL), platelet count ≥ 100 x 109/L (100,000/μL), independent of red cell transfusions for ≥ 1 week immediately before each response assessment. CRh is defined as Response of bone marrow blast <5% with absolute neutrophil count (ANC) > 0.5 × 10^9/L and platelet > 50 × 10^9/L.
Time Frame: From first dose to end of study
Reporting Status: Not Posted, anticipated posting 2026-09

26. Secondary Outcome: Time to Sponsor Derived CR and CRh: Phase 2 (Randomized Phase)
Description: Time from first dose of study drug to first documented CR/CRh. Morphologic Complete Remission (CR) is defined as as less than 5% blasts in a BM aspirate sample with marrow spicules and with a count of at least 200 nucleated cells. There should be no blasts with Auer rods and absence of extramedullary disease. Plus, all the following conditions should be met: ANC ≥ 1 x 109/L (1,000/μL), platelet count ≥ 100 x 109/L (100,000/μL), independent of red cell transfusions for ≥ 1 week immediately before each response assessment. Morphologic complete remission with partial hematologic recovery (CRh) is defined as less than 5% blasts in a BM aspirate sample with marrow spicules plus ANC > 500 x 109/L (1,000/μL) & Platelet count > 50 x 109/L (100,000/μL).
Time Frame: From first dose to end of study
Reporting Status: Not Posted, anticipated posting 2026-09

27. Secondary Outcome: Duration of Sponsor Derived CR/CRh: Phase 2 (Randomized Stage)
Description: Time from first documented CR/CRh to documented morphologic relapse, PD, or death due to any cause, whichever occurred first. Participants without morphologic relapse, PD, or death due to any cause were censored at the date of the last response assessment. Morphologic Relapse is defined as either reappearance of ≥ 5% blasts in the BM not attributable to any other cause or the development of extramedullary disease. Progression (PD) is defined as a > 50% increase of BM blast count percentage from baseline to ≥ 20% for participants with 5 to 70% BM blasts at baseline or a doubling of absolute blast count in peripheral blood from baseline to ≥ 10 x 109/L (10,000/μL) for participants with > 70% BM blasts at baseline or the development of new extramedullary disease.
Time Frame: From first dose to end of study
Reporting Status: Not Posted, anticipated posting 2026-09

ADVERSE EVENTS:
Time Frame: From first dose up to approximately 26 Months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA | Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA | Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA | Phase 1b Expansion Stage: AG-120 (500mg) + AZA | Phase 2 Randomized Stage: AG-221 (100mg) + AZA | Phase 2 Randomized Stage: AZA Monotherapy
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 1/7 | 6/16 | 29/68 | 14/33
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 4/7 | 11/16 | 64/68 | 25/32
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7 | 16/16 | 67/68 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA (N=3) | Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA (N=3) | Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA (N=7) | Phase 1b Expansion Stage: AG-120 (500mg) + AZA (N=16) | Phase 2 Randomized Stage: AG-221 (100mg) + AZA (N=68) | Phase 2 Randomized Stage: AZA Monotherapy (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 7 | 26 | 8
Hyperfibrinolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 0
Catheter site thrombosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Medical device site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 3 | 4 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 1
Chest wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Colonic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cystitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Haemophilus sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Injection site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 2 | 7 | 3
Neutropenic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 0 | 7 | 5
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Scrotal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 2 | 8 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Serratia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Superinfection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Hyphaema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 7 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 3 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 4 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Dose-finding Stage: AG-221 (100mg) + AZA (N=3) | Phase 1b Dose-finding Stage: AG-221 (200mg) + AZA (N=3) | Phase 1b Dose-finding Stage: AG-120 (500mg) + AZA (N=7) | Phase 1b Expansion Stage: AG-120 (500mg) + AZA (N=16) | Phase 2 Randomized Stage: AG-221 (100mg) + AZA (N=68) | Phase 2 Randomized Stage: AZA Monotherapy (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 7 | 35 | 15
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 3 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 6 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 6 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 5 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 3 | 31 | 9
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 5 | 7 | 40 | 14
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 2 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | 3 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 4 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 4 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 1 | 3 | 1
Lacrimation decreased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 2 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 3 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 0 | 4 | 12 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 4 | 7 | 31 | 15
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 5 | 9 | 29 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 4 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 6 | 8 | 47 | 12
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 10 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 9 | 33 | 11
Asthenia (General disorders) | 0 | 1 | 0 | 3 | 16 | 4
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 3 | 2
Chills (General disorders) | 0 | 0 | 1 | 1 | 4 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 5 | 4 | 19 | 8
Gait disturbance (General disorders) | 1 | 1 | 0 | 0 | 1 | 0
Granuloma (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infusion site discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 2 | 3 | 11 | 7
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site irritation (General disorders) | 0 | 0 | 1 | 0 | 0 | 2
Injection site pain (General disorders) | 0 | 0 | 0 | 2 | 2 | 3
Injection site pruritus (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Injection site reaction (General disorders) | 0 | 1 | 0 | 1 | 3 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 3
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 2 | 6 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1 | 4 | 20 | 10
Pain (General disorders) | 0 | 0 | 0 | 1 | 4 | 2
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 2 | 5 | 19 | 6
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Granulomatous liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 6 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Immunodeficiency (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 6 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 2
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 3 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 5 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 11 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 1 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 2 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 3 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 2
Amylase increased (Investigations) | 0 | 0 | 2 | 0 | 2 | 1
Antithrombin III decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 5 | 3
Blood bilirubin increased (Investigations) | 1 | 3 | 1 | 1 | 19 | 1
Blood chloride decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 4 | 3
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Carbon dioxide increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 7 | 6 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 5 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 1 | 2 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 2 | 2 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2 | 3 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 6 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 0 | 2 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 5 | 25 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 5 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 7 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 5 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 6 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 5 | 25 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 6 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 5 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 10 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 6 | 12 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 5 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 8 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 2
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 6 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 3 | 3 | 17 | 3
Dysgeusia (Nervous system disorders) | 2 | 1 | 0 | 2 | 5 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 4 | 14 | 5
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 4 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 0
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 2 | 8 | 3
Claustrophobia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 2 | 3 | 1
Delirium (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 3 | 4 | 3
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 4 | 13 | 3
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 2 | 1 | 11 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 3 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 3 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 1
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 4 | 13 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 13 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 12 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 4 | 2
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 3 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 3 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 3 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 8 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1
Aortic thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 4 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 5 | 3
Hypotension (Vascular disorders) | 2 | 1 | 1 | 2 | 13 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT02677922/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT02677922/SAP_001.pdf